CLINICAL TRIAL: NCT03394417
Title: StrataXRT vs Standard Clinical Practice for the Prevention of Acute Dermatitis in Patients Receiving Concurrent Chemoradiation for Head and Neck Cancers
Brief Title: StrataXRT vs Standard Clinical Practice for the Prevention of Acute Dermatitis in Head and Neck Cancers Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016/01084
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancers; Acute Radiation Dermatitis
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard clinical practice (control) (No Intervention): aqueous cream normally prescribed by radiation oncologists
- StrataXRT (intervention) (Active Comparator): silicon-based gel for radiation dermatitis
  Interventions: Device: StrataXRT

INTERVENTIONS:
Device: StrataXRT — randomized patient allocated to this group will receive StrataXRT for application during the treatment and 4 weeks further after the treatment ends.
  Arms: StrataXRT (intervention)

SUMMARY:
This is a phase IV, prospective, double-blind, randomized controlled trial with 2 study arms. The study population will be patients receiving chemoradiation for head and neck carcinomas, the majority of whom will be outpatients unless they require inpatient supportive care during treatment.

There will be a 12 to 14-week longitudinal follow-up with 9 assessments conducted during this follow-up.

The estimated duration of recruitment will be 6-8 years.

Intervention group If a patient is allocated to the intervention group following randomization, the patient will be treated with StrataXRT.

Control group If a patient is allocated to the control group following randomization, the patient will be treated with standard clinical practice which consists of aqueous cream.

DETAILED DESCRIPTION:
Clinical significance and current evidence:

Radiation dermatitis occurs commonly in patients receiving chemoradiation for nasopharyngeal cancer; 50 to 60% develop grade 2 or higher dermatitis. This can result in significant morbidity, reduced aesthetic appearance, decrease in quality of life and delays in treatment. Current literature does not conclusively support the use of one agent over another for prevention of radiation dermatitis. The choice of agents used in clinical practice is highly variable, with aqueous agents being one of the commonest.

Specific Aims:

The aim of this study is to evaluate if the investigational product (StrataXRT), a silicone-based gel, is superior to standard clinical practice in prevention of grade 2 or higher acute dermatitis in patients receiving chemoradiation for nasopharyngeal carcinoma.

Trial Design:

The study will be conducted using a prospective, double-blind randomized control trial in 2 institutions. Each arm will receive standard radiation to a total dose of 70 Gray (Gy) with concurrent chemotherapy. The primary objective is to compare the prevention of dermatitis and the primary endpoint is reached when grade 2 or higher dermatitis according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 scale occurs. Secondary objectives will be evaluation of the time to onset of dermatitis, the time to complete recovery from dermatitis and the degree of pain. Assessment of the patient's skin will be done at baseline, weekly during treatment, 1 week post treatment and unless the skin has resolved to baseline then every week up until 6 weeks post-treatment, which will mark the end of follow-up. The safety end-point is reached when grade 4 dermatitis occurs.

Hypothesis and statistics:

The investigators aim to demonstrate a 30% reduction in the incidence of grade 2 or higher dermatitis with StrataXRT. Using a 2-sided test at significance level 0.05 to detect the difference with a power of 80%, the investigators envisage a recruitment of 100-150 patients in total. The study duration is estimated to be 8 years.

ELIGIBILITY:
Inclusion Criteria:

* patients who are 21 years of age or older
* histological diagnosis of head and neck carcinoma available
* patients who are to be treated with concurrent chemoradiation
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3
* no known allergy to StrataXRT or silicone
* able to give written informed consent, or have written consent given on their behalf

Exclusion Criteria:

* patients who cannot apply the skin product or have it administered to them
* patients with comorbidities and/or on medications that may alter the response of the skin e.g. connective tissue disorder
* patients with existing rashes or wounds in the radiation field at baseline
* patients receiving concurrent cetuximab during radiotherapy
* previous radiotherapy to the head and neck region
* female patients who are pregnant or breast feeding
* unable to give written informed consent , or are unable to have written consent given on their behalf

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
grade 2 acute radiation dermatitis | 10 weeks
  when patient develops grade 2 acute radiation dermatitis as scored by Common Terminology Criteria for Adverse Event (CTCAE) version 4.03 scale with grade 1 the mildest, Grade 1: faint erythema or dry desquamation Grade 2: moderate to brisk erythema; patchy moist desquamation; moderate edema Grade 3: moist desquamation other than skin folds and creases; bleeding induced by minor trauma or abrasion Grade 4: skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site Grade 5: death

SECONDARY OUTCOMES:
completion of scheduled post-treatment assessment at 6 weeks post-radiotherapy | 12 weeks
  when patient completed the scheduled post-radiotherapy assessment

CONTACTS AND LOCATIONS:
Overall Officials: David Chia, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided